CLINICAL TRIAL: NCT06184165
Title: Stratifying Psychoses for Personalized REpetitive TMS in Persistent NEgative Symptoms Alleviation
Acronym: SP-RENESA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8371
Record Dates: First submitted 2023-11-20; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Persistent Negative Symptoms; Progressive Periodic Catatonia; Aviation; Apathy
MeSH Terms: conditions — Schizophrenia; Lethargy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Informants (caregivers)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- N°1: PMI in PPC (Experimental): Progressive periodic catatonia (SSD phenotype) Premotor inhibition using personalized rTMS (40 sec continuous theta-burst on each of the 5 targets corresponding to hyper-perfused regions, i.e. functional biomarker, 120%).
  N = 40.
  Interventions: Procedure: Personalized rTMS
- N°2: PFA in PPC (Active Comparator): Progressive periodic catatonia (SSD phenotype) Classical left-prefrontal activation using intermittent theta-burst rTMS (72 trains, 120%).
  N = 40.
  Interventions: Procedure: Personalized rTMS
- N°3: PMI in nPPC (Active Comparator): Other phenotype of SSD than PPC (nPPC) Premotor inhibition using personalized rTMS (40 sec continuous theta-burst on each of the 5 targets corresponding to most perfused premotor regions).
  N = 40.
  Interventions: Procedure: Personalized rTMS
- N°4: PFA in nPPC (Experimental): Non-progressive periodic catatonia SSD phenotype Classical left-prefrontal activation (PFA) using intermittent theta-burst rTMS (72 trains, 120%).
  N = 40.
  Interventions: Procedure: Personalized rTMS

INTERVENTIONS:
Procedure: Personalized rTMS — 5 "personalized" targets accessible to TMS (at less than 3.5 cm distance from the scalp or the coil's hot spot) are placed in the hyper-perfused premotor regions.
  The patient is installed on the robotic device. The technician puts a neuro-navigation tracker on the subject's forehead and proceeds to the co-registration. The motor threshold is defined, and stimulator output's intensity is adjusted accordingly (120%) The robotic system ensures that the actual stimulation is performed according to the personalized protocol. This adequacy will be evaluated secondarily based on the recordings of the coil positions during each

SUMMARY:
In its 2012's release guideline on therapy for schizophrenia, the EMA joined the FDA to acknowledge primary and persistent negative symptoms (PNS) as an unmet need in the treatment of schizophrenia. Functional brain imaging studies showed a correlation between NS and reduced perfusion in the left dorsolateral prefrontal cortex (L-DLPFC). Pre-frontal activation (PFA) using repetitive transcranial magnetic stimulation (rTMS) significantly improve PNS (meta-analyses: effect size SMD = 0.55, ΔPANSS-N = -2.5). Yet schizophrenia is likely to gather many different natural entities of distinct pathophysiological mechanisms. Pursuing a one-size-fits-all approach will not adapt to this diversity and might account for inconsistencies in the results.

Progressive periodic catatonia (PPC) is a rare psychotic phenotype (0.1 - 0.5 ‰) which has been shown to be longitudinally stable (30-years follow-up) and consistent within families (about 1 third of first-degree relatives are affected). The core of this phenotype is a disintegration of psychomotor processes which progresses with each relapse, resulting in a "deficit state", i.e., PNS, responsible for most social and occupational disabilities. The investigators and others reported PPC to come with hyper-perfusions in premotor cortices compared to controls or non-PPC chronic psychoses (nPPC). These hyper-perfusions discriminate PPC from nPPC or depressive patients (Sensitivity = 82%; Specificity = 95%). Last, in independent proof-of-principle studies the investigators and others have shown that premotor inhibition (PMI) using rTMS significantly improved PNS in PPC and that the most dramatic improvements followed personalized accelerated rTMS protocols (5 days of rTMS; CGI-improvement = 2 which is equivalent to ΔPANSS-N = -10; lasting > 1 month - vs virtually no change for PFA). The efficacy index was very good (no side effects).

the investigators hypothesize that: (1) in PPC, add-on personalized premotor inhibition (PMI) is more effective in reducing PNS than L-DLPFC activation (PFA); (2) patient stratification is relevant as personalized PMI will not be as effective in the nPPC group (even expected to be less effective than PFA).

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age; affiliated to health insurance; superior or equal to B2 level of linguistic competency in French.
* Suffering from schizophrenia spectrum disorder (SSD) in residual state with persistent negative symptoms (PNS): (1) SSD: ICD-11 codes beginning with 6A2 + primary catatonia (codes beginning with 6A4) + simple schizophrenia as defined in ICD-10 (F20.6); (2) PNS: persistence (≥6 months - based on patient ± informant's interview) of ≥2 negative symptoms (PANSS-N1, N2, N3, N4, N6 ≥4) with functional impact.
* Half of subjects having PPC, the other half suffering from another phenotype or nPPC (neuropsychiatric procedure or probabilistic, i.e. Bayes-PPC).
* Under a stable medication regimen for >6 weeks,
* Subjects who have received the protocol information and signed informed consent.

Exclusion Criteria:

* - Contraindications for MRI or rTMS.
* Motor deficit at neurological examination.
* Secondary negative symptoms: (1) withdrawal secondary to severe anxiety (especially due to positive symptoms), (2) depression, (3) maintenance on high dose antipsychotics, (4) extra-pyramidal or (5) sedation side-effects, (6) treatment non-compliance, (7) current substance abuse (except nicotine and caffeine), (8) unsubstituted past opioid addiction, (9) poor health or social condition.
* Under antiepileptic drugs (except lamotrigine and long-term use of benzodiazepines).
* Pregnancy; severe medical condition; care under constraint.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Decrement in positive and negative syndrome scale - negative sub-score (ΔPANSS-N). | Pre-rTMS and end-of-trial (before - week 4, and 6 weeks after rTMS - week12).
  Positive and negative syndrome scale - negative sub-score ΔPANSS-N = ΔN1 + ΔN2 + ΔN3 + ΔN4 + ΔN6
  PMI personalized rTMS superiority claim in PPC: ANOVA within-between 2 factors interaction (two-way comparison):
  * The within factor is "pre-rTMS/end-of-study", i.e., PNS change between the 2 repeated measures: PANSS-N before and at 1.5-months after rTMS.
  * The between factor is "treatment arm": PMI vs PFA.
  Precision medicine claim (phenotype-dependent response): 3-way ANOVA (interaction between the 2 between and 1 within factors):
  * The within factor is "pre/end", i.e., PNS change between the 2 repeated measures: PANSS-N before and at 1.5-months after rTMS.
  * The first between factor is "treatment arm": PMI vs PFA.
  * The second between factor is "phenotype": PPC vs nPPC.

IPD SHARING:
Plan to Share IPD: No